CLINICAL TRIAL: NCT00948389
Title: Randomized Phase II of Lomustine Versus Lomustine-Dasatinib in Patients With Recurrent Glioblastoma
Brief Title: Study of CCNU (Lomustine) Plus Dasatinib in Recurrent Glioblastoma (GBM)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Inability to meet protocol objectives
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA180-274; Protocol 26083 (Other: EORTC); 2009-010576-21 (EudraCT Number)
Record Dates: First submitted 2009-07-28; First posted 2009-07-29 (Estimated); Results first posted 2012-08-28 (Estimated); Last update posted 2012-08-31 (Estimated); Status verified 2012-08

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Dasatinib; Lomustine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dasatinib (Active Comparator)
  Interventions: Drug: Dasatinib
- Lomustine (Active Comparator)
  Interventions: Drug: Lomustine

INTERVENTIONS:
Drug: Dasatinib — Tablets, Oral, 100 mg, Once or Twice daily (depending on safety cohort), Until progression or toxicity
  Other Names: BMS-354825
  Arms: Dasatinib
Drug: Lomustine — Tablets, Oral, 110 mg/m², Every 6 weeks, until progression or toxicity
  Arms: Lomustine

SUMMARY:
To determine whether dasatinib plus lomustine are effective for treatment of recurrent glioblastoma

ELIGIBILITY:
Inclusion Criteria:

* Patients with histological or cytological proven glioblastoma multiforme
* Recurrent or progressive disease documented by magnetic resonance imaging (MRI)
* World Health Organization (WHO) Performance status 0 - 2
* Patient may have been operated for recurrence
* For non operated patients, recurrent disease must be at least one bidimensionally measurable target lesion with one diameter of at least 2cm
* Patients must be on a stable or decreasing dose of corticosteroids for at least 1 week prior to baseline MRI

Exclusion Criteria:

* Patients with histological or cytological proven glioblastoma multiforme
* Completion of radiotherapy to the brain less than 3 months prior to registration/randomization
* Prior treatment with high dose radiotherapy, stereotactic radiosurgery or internal radiation therapy
* Previous or current malignancy at other sites within prior 3 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2009-10; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (5):
- Local Institution, Paris, France
- Local Institution, Bologna, Italy
- Netherlands (2):
  - Local Institution, Nijmegen
  - Local Institution, Rotterdam
- Local Institution, Lausanne, Switzerland

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 28 participants enrolled in this study, 26 received treatment.
Groups:
- Dasatinib, 100 mg QD/100 mg BID + Lomustine, 110 mg/m^2: Dose level 1A. Cycle 1: Dasatinib, 100 mg once daily (QD). Cycle 2: Dasatinib, 100 mg twice daily (BID), plus lomustine, 110 mg/m^2.
- Dasatinib, 100 mg QD/100 mg BID + Lomustine, 90 mg/m^2: Dose level 1B. Cycle 1: Dasatinib,100 mg QD. Cycle 2: 100 mg BID, plus lomustine, 90 mg/m^2.
- Dasatinib, 100 mg BID + Lomustine, 90 mg/m^2: Dose level 2. Dasatinib, 100 mg BID plus lomustine, 90 mg/m^2
- Dasatinib, 150 mg/d + Lomustine, 90 mg/m^2: Dose level 3A: Dasatinib, 150 mg/d (100 mg AM and 50 mg PM), plus lomustine, 90 mg/m^2
- Dasatinib, 100 mg/d QD + Lomustine, 90 mg/m^2: Dose Level 3B: Dasatinib, 100 mg/d QD plus lomustine, 90 mg/m^2
Period: Overall Study
Arm/Group | Dasatinib, 100 mg QD/100 mg BID + Lomustine, 110 mg/m^2 | Dasatinib, 100 mg QD/100 mg BID + Lomustine, 90 mg/m^2 | Dasatinib, 100 mg BID + Lomustine, 90 mg/m^2 | Dasatinib, 150 mg/d + Lomustine, 90 mg/m^2 | Dasatinib, 100 mg/d QD + Lomustine, 90 mg/m^2
Started | 6 | 3 | 7 | 9 | 1
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 6 | 3 | 7 | 9 | 1
Not completed — Disease Progression/Relapse/Death | 3 | 3 | 7 | 8 | 1
Not completed — Thrombocytopenia, Grade 4 | 2 | 0 | 0 | 1 | 0
Not completed — Both Progression and Toxicity | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Dose Level 1A: Dasatinib: 100 mg once daily (QD) cycle 1 / 100 mg twice daily (BID) cycle 2 + lomustine (CCNU): 110 mg/m²
- Dose Level 1B: Dasatinib: 100 mg QD / 100mg BID + CCNU: 90 mg/m²
- Dose Level 2: Dasatinib: 100 mg BID + CCNU: 90 mg/m²
- Dose Level 3A: Dasatinib: 150 mg/day (100 mg AM and 50 mg PM) + CCNU: 90 mg/m²
- Dose Level 3B: Dasatinib: 100 mg/day (QD) + CCNU: 90 mg/m²
- Total: Total of all reporting groups
Arm/Group | Dose Level 1A | Dose Level 1B | Dose Level 2 | Dose Level 3A | Dose Level 3B | Total
Number analyzed (Participants) | 6 | 3 | 7 | 9 | 1 | 26
Age Continuous [Median (Full Range); unit: years] | 58.8 [41.3 to 70.7] | 57.7 [48.9 to 57.7] | 53.6 [42.4 to 64.0] | 49.7 [38.8 to 66.8] | 51.1 [51.1 to 51.1] | 54.8 [38.8 to 70.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 2 | 3 | 0 | 6
  Male | 5 | 3 | 5 | 6 | 1 | 20
Histological Diagnosis of Primary Disease [Number; unit: participants] — by local pathologist
  participants
    glioblastoma multiforme | 6 | 2 | 5 | 8 | 1 | 22
    glioblastoma w/ oligodendroglial component | 0 | 1 | 2 | 1 | 0 | 4
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — ECOG criteria is used to assess disease progression and affects on daily living abilities and to determine appropriate treatment and prognosis. Grade 0=normal activity; Grade 1=Restricted physical activity but ambulatory and capable of light work; Grade 2=Ambulatory, capable of self care, but unable to carry out any work activities; Grade 3=Capable of limited self care, confined to bed or chair 50% or more of waking hours; Grade 4=Completely disabled, totally confined to bed or chair.
  participants
    Grade 0 | 6 | 2 | 1 | 4 | 1 | 14
    Grade 1 | 0 | 1 | 5 | 4 | 0 | 10
    Grade 2 | 0 | 0 | 1 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs), Serious AEs (SAEs), Deaths, and Discontinuations Due to AEs
Description: SAE=any untoward medical event that results in death, persistent or significant disability/incapacity, or drug dependency or abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires inpatient hospitalization or prolongation. AE=any new untoward medical occurrence or worsening of a preexisting medical condition that does not necessarily have a causal relationship with this treatment. Treatment-related(Tx-R)=certainly, probably, possibly related and unknown relationship to study drug. AE grades(Gr) 1=Mild; 2=Moderate; 3=Severe; 4=Life-threatening.
Time Frame: Assessed at baseline, every 2 weeks during cycles 1-6 (6-week cycles), and every 6 weeks after cycle 6. Median number of cycles = 1.0 (range: 1.0 - 7.0).
Population: All treated participants
Measure: Number; unit: participants
Arm/Group | Dasatinib, 100 mg QD/100 mg BID + Lomustine, 110 mg/m^2 | Dasatinib, 100 mg QD/100 mg BID + Lomustine, 90 mg/m^2 | Dasatinib, 100 mg BID + Lomustine, 90 mg/m^2 | Dasatinib, 150 mg/d + Lomustine, 90 mg/m^2 | Dasatinib, 100 mg/d QD + Lomustine, 90 mg/m^2
Number analyzed (Participants) | 6 | 3 | 7 | 9 | 1
participants
  Deaths within 30 days of Tx Discontinuation | 1 | 0 | 1 | 0 | 0
  Tx-R Deaths within 30 days of Tx Discontinuation | 0 | 0 | 0 | 0 | 0
  At Least 1 SAE | 5 | 1 | 4 | 4 | 0
  At Least 1 Tx-R SAE | 4 | 0 | 1 | 1 | 0
  Discontinuations Due to AEs | 3 | 0 | 0 | 1 | 0
  At Least 1 AE | 6 | 3 | 7 | 9 | 1
  At Least 1 Gr 3/4 AE | 2 | 2 | 4 | 4 | 0
  At Least 1 Tx-R AE | 5 | 2 | 5 | 7 | 1
  At Least 1 Tx-R Gr 3/4 AE | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Dose-limiting Toxicities (DLTs)
Description: Grades (gr) according to National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI CTCAE), version 3.0. DLTs were defined as adverse drug reactions as follows: absolute neutrophil counts <0.5x10^9/L (gr4) lasting for 7 consecutive days; febrile neutropenia (neutrophil count <1x10^9/L and fever of >=38.5°C); thrombocytopenia (gr4); any gr3/4 nonhematological toxicity except nausea, vomiting and fever which could be rapidly controlled with appropriate measures; any toxicity which did not allow administering at least 70% of the intended dose intensity for both agents.
Time Frame: The duration for observation of DLT was 2 6-week cycles in participants with escalated dose (QD to BID) and 1 6 -week cycle for participants starting with BID regime. For participants receiving dasatinib at 150 mg, DLTs were only documented over cycle 1.
Population: Evaluable Participants: subset of participants used to decide on dose escalations. Participants were assessable if they completed the period for DLT observation.
Measure: Number; unit: participants
Arm/Group | Dasatinib, 100 mg QD/100 mg BID + Lomustine, 110 mg/m^2 | Dasatinib, 100 mg QD/100 mg BID + Lomustine, 90 mg/m^2 | Dasatinib, 100 mg BID + Lomustine, 90 mg/m^2 | Dasatinib, 150 mg/d + Lomustine, 90 mg/m^2 | Dasatinib, 100 mg/d QD + Lomustine, 90 mg/m^2
Number analyzed (Participants) | 5 | 0 | 5 | 9 | 0
participants | 3 |  | 3 | 4 |

3. Primary Outcome: Deaths Within 30 Days of Protocol Treatment Discontinuation
Time Frame: From time of randomization through within 30 days after protocol treatment discontinuation. Median (full range) number of 6-week treatment cycles was 1.0 (1.0-7.0).
Population: Treated participants
Measure: Number; unit: participants
Arm/Group | Dasatinib, 100 mg QD/100 mg BID + Lomustine, 110 mg/m^2 | Dasatinib, 100 mg QD/100 mg BID + Lomustine, 90 mg/m^2 | Dasatinib, 100 mg BID + Lomustine, 90 mg/m^2 | Dasatinib, 150 mg/d + Lomustine, 90 mg/m^2 | Dasatinib, 100 mg/d QD + Lomustine, 90 mg/m^2
Number analyzed (Participants) | 6 | 3 | 7 | 9 | 1
participants | 1 | 0 | 1 | 0 | 0

4. Primary Outcome: Number of Participants With Worst Grade of Hematological Toxicity Per NCI CTCAE Version 3.0 Criteria
Description: Neutrophils (neutropenia): Grade (gr)1 <LLN-1500/mm3; Gr2 <1500-1000/mm3; Gr3 <1000-500/mm3; Gr4 <500/mm3. Leukocytes (leukopenia): Gr1 <LLN-3000/mm3; Gr2 <3000-2000/mm3; Gr3 <2000-1000/mm3; Gr4 <1000/mm3. Lymphocytes (lymphocytopenia): Gr1 <LLN-800/mm3; Gr2 <800-500/mm3; Gr3 <500-200/mm3; Gr4 <200/mm3. Platelets (thrombocytopenia): Gr1 <LLN-75,000/mm3; Gr2 <75,000-50,000/mm3; Gr3 <50,000-25,000/mm3; Gr4 <25,000/mm3. Hemoglobin (anemia): Gr1 <LLN-10.0 g/dL; Gr2 <10.0-8.0 g/dL; Gr3 <8.0-6.5 g/dL; Gr4 <6.5 g/dL. LLN/ULN=lower/upper limit of normal (normal ranges may vary by local laboratories).
Time Frame: as for outcome 1
Population: Treated participants
Measure: Number; unit: participants
Arm/Group | Dasatinib, 100 mg QD/100 mg BID + Lomustine, 110 mg/m^2 | Dasatinib, 100 mg QD/100 mg BID + Lomustine, 90 mg/m^2 | Dasatinib, 100 mg BID + Lomustine, 90 mg/m^2 | Dasatinib, 150 mg/d + Lomustine, 90 mg/m^2 | Dasatinib, 100 mg/d QD + Lomustine, 90 mg/m^2
Number analyzed (Participants) | 6 | 3 | 7 | 9 | 1
participants
  At least 1 Grade 1-4 Neutropenia | 3 | 2 | 2 | 5 | 0
  At least 1 Grade 1-4 Leukopenia | 5 | 3 | 4 | 6 | 0
  At least 1 Grade 1-4 Lymphocytopenia | 5 | 2 | 4 | 9 | 0
  At least 1 Grade 1-4 Thrombocytopenia | 6 | 3 | 6 | 9 | 1
  At least 1 Grade 1-4 Anemia | 6 | 1 | 6 | 9 | 0
  At least 1 Grade 3-4 Neutropenia | 2 | 1 | 0 | 4 | 0
  At least 1 Grade 3-4 Leukopenia | 1 | 1 | 0 | 4 | 0
  At least 1 Grade 3-4 Lymphocytopenia | 4 | 0 | 1 | 5 | 0
  At least 1 Grade 3-4 Thrombocytopenia | 4 | 0 | 2 | 5 | 0
  At least 1 Grade 3-4 Anemia | 0 | 0 | 1 | 0 | 0

5. Primary Outcome: Number of Participants With Worst Grade of Biochemistry Abnormality Per NCI CTCAE Version 3.0 Criteria
Description: Grades (gr) 1=mild; gr2=moderate; gr3=severe; gr4=life-threatening. For details of NCI CTCAE laboratory values for each grade, please refer to http://ctep.cancer.gov/protocolDevelopment/electronic_applications/ctc.htm#ctc_30. Low Potassium=Hypokalemia, High Potassium=Hyperkalemia, Low Sodium=Hyponatremia, Low Calcium=Hypocalcemia, High Bilirubin=Hyperbilirubinemia, low phosphatase=Hypophosphatemia, Low Potassium=Hypokalemia.
Time Frame: Assessed at baseline, every 2 weeks during cycles 1-6 (6-week cycles), and every 6 weeks after 6 cycles. Median number of cycles = 1.0 (range: 1.0 - 7.0).
Population: Treated participants
Measure: Number; unit: participants
Arm/Group | Dasatinib, 100 mg QD/100 mg BID + Lomustine, 110 mg/m^2 | Dasatinib, 100 mg QD/100 mg BID + Lomustine, 90 mg/m^2 | Dasatinib, 100 mg BID + Lomustine, 90 mg/m^2 | Dasatinib, 150 mg/d + Lomustine, 90 mg/m^2 | Dasatinib, 100 mg/d QD + Lomustine, 90 mg/m^2
Number analyzed (Participants) | 6 | 3 | 7 | 9 | 1
participants
  At least 1 Gr 1-4 Hypokalemia | 1 | 0 | 1 | 3 | 0
  At least 1 Gr 1-4 Hyperkalemia | 0 | 1 | 0 | 0 | 0
  At least 1 Gr 1-4 Hyponatremia | 1 | 0 | 0 | 0 | 0
  At least 1 Gr 1-4 Hypernatremia | 1 | 1 | 0 | 5 | 0
  At least 1 Gr 1-4 Creatinine | 0 | 2 | 0 | 0 | 0
  At least 1 Gr 1-4 Hypocalcemia | 3 | 1 | 3 | 2 | 0
  At least 1 Gr1-4 Hyperbilirubinemia | 0 | 0 | 0 | 0 | 1
  At least 1 Gr 1-4 Aspartate Aminotransferase / AST | 2 | 0 | 4 | 6 | 0
  At least 1 Gr 1-4 Hypophosphatemia | 1 | 1 | 1 | 3 | 0
  At least 1 Gr 3-4 Hypokalemia | 0 | 0 | 0 | 1 | 0

6. Other Pre Specified Outcome: Number of Participants With Disease Progression at 12 Months
Description: As measured by brain magnetic resonance imaging.
Time Frame: 12 months
Population: Treated participants
Measure: Number; unit: participants
Arm/Group | Dasatinib, 100 mg QD/100 mg BID + Lomustine, 110 mg/m^2 | Dasatinib, 100 mg QD/100 mg BID + Lomustine, 90 mg/m^2 | Dasatinib, 100 mg BID + Lomustine, 90 mg/m^2 | Dasatinib, 150 mg/d + Lomustine, 90 mg/m^2 | Dasatinib, 100 mg/d QD + Lomustine, 90 mg/m^2
Number analyzed (Participants) | 6 | 3 | 7 | 9 | 1
participants | 6 | 3 | 7 | 9 | 1

ADVERSE EVENTS:
Arm/Group | Dasatinib, 100 mg QD/100 mg BID + Lomustine, 110 mg/m^2 | Dasatinib, 100 mg QD/100 mg BID + Lomustine, 90 mg/m^2 | Dasatinib, 100 mg BID + Lomustine, 90 mg/m^2 | Dasatinib, 150 mg/d + Lomustine, 90 mg/m^2 | Dasatinib, 100 mg/d QD + Lomustine, 90 mg/m^2
Serious Adverse Events (participants affected / at risk) | 5/6 | 1/3 | 4/7 | 3/9 | 0/1
Other Adverse Events (participants affected / at risk) | 6/6 | 3/3 | 7/7 | 9/9 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dasatinib, 100 mg QD/100 mg BID + Lomustine, 110 mg/m^2 (N=6) | Dasatinib, 100 mg QD/100 mg BID + Lomustine, 90 mg/m^2 (N=3) | Dasatinib, 100 mg BID + Lomustine, 90 mg/m^2 (N=7) | Dasatinib, 150 mg/d + Lomustine, 90 mg/m^2 (N=9) | Dasatinib, 100 mg/d QD + Lomustine, 90 mg/m^2 (N=1)
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 1 | 1 | 2 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 2 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Enteritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Death (General disorders) | 1 | 0 | 1 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Brain oedema (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Platelet count decreased (Investigations) | 2 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dasatinib, 100 mg QD/100 mg BID + Lomustine, 110 mg/m^2 (N=6) | Dasatinib, 100 mg QD/100 mg BID + Lomustine, 90 mg/m^2 (N=3) | Dasatinib, 100 mg BID + Lomustine, 90 mg/m^2 (N=7) | Dasatinib, 150 mg/d + Lomustine, 90 mg/m^2 (N=9) | Dasatinib, 100 mg/d QD + Lomustine, 90 mg/m^2 (N=1)
Agitation (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 1 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0 | 0
Prostatism (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Speech disorder (Nervous system disorders) | 1 | 2 | 1 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 1 | 0
Carbon monoxide diffusing capacity (Investigations) | 0 | 2 | 3 | 3 | 1
Convulsion (Nervous system disorders) | 0 | 1 | 0 | 1 | 0
Cystitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Ocular surface disease (Eye disorders) | 0 | 0 | 1 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 4 | 1 | 3 | 5 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Conduction disorder (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 1 | 2 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Hemianopia homonymous (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 4 | 1 | 4 | 6 | 0
Peripheral coldness (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 2 | 2 | 1 | 0
Urethral haemorrhage (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Weight increased (Investigations) | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Dry eye (Eye disorders) | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 3 | 1 | 4 | 3 | 1
Memory impairment (Nervous system disorders) | 0 | 1 | 1 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Skin infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0
Adverse event (General disorders) | 0 | 0 | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 6 | 3 | 6 | 6 | 1
Pollakiuria (Renal and urinary disorders) | 3 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 4 | 0 | 3 | 5 | 1
Weight decreased (Investigations) | 1 | 1 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Hemianopia (Nervous system disorders) | 0 | 0 | 0 | 2 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0 | 0
Optic neuropathy (Eye disorders) | 2 | 0 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Brain oedema (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Depressed mood (Psychiatric disorders) | 0 | 2 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 4 | 3 | 0
Face oedema (General disorders) | 1 | 0 | 0 | 0 | 0
Hyperaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Neoplasm swelling (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 3 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 1 | 2 | 0
Exfoliative rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Penile ulceration (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.